CLINICAL TRIAL: NCT06717308
Title: Surgical Drape With an Atraumatic Acrylic Adhesive for Negative Pressure Wound Therapy
Brief Title: Evaluation of a Switchable Acrylic Adhesive Drape for Safer Removal in Negative Pressure Wound Therapy Applications.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Global Biomedical Technologies, LLC (Industry)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Weill Medical College of Cornell University (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R44EB036280 (NIH); 1R44EB036280-01 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2024-12-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Frequency and Type of Medical Adhesive-Related Skin Injury; NPWT Drape Seal Effectiveness Rate (or Leak Incidence Rate); Clinician Acceptability of New NPWT Drape; Patient Drop-out Rate From Prescribed NPWT Treatment; Pain Assessment During Medical Adhesive Drape Removal
Keywords: Medical Adhesive-Related Skin Injury (MARSI); pain with adhesive medical products; wound care; NPWT drape; Negative Pressure Wound Therapy; Surgical Drapes

STUDY DESIGN:
Intervention Model Description: 50% of the patients will receive the KCI® drape (control), and 50% of the patients will receive the Comfort Release® drape (intervention). Outcomes assessed will include the effectiveness of the seal, pain during dressing removal, skin damage upon removal, and clinician acceptability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Single use post surgical NPWT drape application (Active Comparator): Aim 1 description: A comparison of performance of Comfort Release® drapes with V.A.C. drapes in single-use NPWT applications in a randomized controlled trial. Post-surgical patients (n=200) with a prescribed treatment of Negative Pressure Wound Therapy (NPWT), will be enrolled at Weill Cornell under PI. Dr. Robert Winchell and at Columbia Presbyterian hospital under co-Principal Investigator Dr. Jarrod Bogue, and Absolute Medical Center under PI: Daniel Careage, MD, for single-use NPWT. Patients will be randomized to a single use control (V.A.C. drape) or intervention (Comfort Release® drape). All other components of the NPWT device including but not limited to the pump, tubing, foam or dressing insert and will be identical. Randomize patients- 1/2 of the patients to receive KCI drape and 1/2 to receive the intervention - Comfort Release drape. The intervention is a change in a component in the NPWT treatment kit.
  Interventions: Device: Comfort Release® NPWT drape
- Multi-use chronic wound NPWT drape application (Active Comparator): Aim 2: A comparison of the performance of Comfort Release® drapes with V.A.C. drapes in serial-use NPWT applications in a randomized controlled trial. Chronic wound patients (n=100) with prescribed NPWT will be enrolled at Weill Cornell Medical Center under Principal Investigator Dr. Robert Winchell and Vital Medical Research under Deeza Frankel, DPM. All patients will undergo 3 NPWT drape changes per week. Patients will be randomized to control (V.A.C. drape.) or intervention (Comfort Release® drape) for the duration of their study enrollment. All other components of the NPWT device including but not limited to the pump, tubing, foam or dressing insert will be identical.
  Randomize patients- 1/2 of the patients to receive KCI drape and 1/2 to receive the intervention- Comfort Release drape. The intervention is a change in a component in the NPWT treatment kit.
  Interventions: Device: Comfort Release® NPWT drape

INTERVENTIONS:
Device: Comfort Release® NPWT drape — Comfort Release® NPWT drape- painless and trauma-free removal, as compared to the control NPWT drape.

SUMMARY:
Negative pressure wound therapy (NPWT) is widely used for chronic and acute wounds, severe burns, and post-operative care. Despite its benefits, the strong adhesive required to maintain an airtight seal increases the risk of medical adhesive-related skin injuries (MARSI), pain, and discomfort during removal. Global Biomedical Technologies (GBT) aims to develop an NPWT drape with "switchable adhesive" technology to enhance removal while maintaining an effective seal. This innovation is expected to benefit both single-use and serial-use NPWT applications by reducing MARSI and improving patient comfort.

This project will compare the functionality and acceptability of Comfort Release® NPWT drapes with the industry-standard V.A.C. drape (KCI Technologies, Inc.) in a non-blinded randomized controlled trial.

Specific Aims Aim 1: Compare Comfort Release® drapes with V.A.C. drapes in single-use NPWT applications in post-surgical patients (n=200) at Columbia University Medical Center, Weill Cornell Medical Center, and Absolute Medical Center.

Milestones: Demonstrate statistically significant (α=0.05) improvement over V.A.C. drapes in:

Reduction of MARSI (Medical Adhesive-Related Skin Injury scoring system) Decreased pain (Indiana Polyclinic Combined Pain Scale) Reduced need for pain/anxiety medication Equivalent or improved seal effectiveness (leak incidence rate) Clinician acceptability Aim 2: Compare Comfort Release® drapes with V.A.C. drapes in serial-use NPWT applications in chronic wound patients (n=100) at Weill Cornell Medical Center and Vital Medical Research. Patients will undergo three NPWT drape changes per week.

Milestones: Demonstrate statistically significant (α=0.05) improvement over V.A.C. drapes in:

Reduction of MARSI Decreased pain (Indiana Polyclinic Combined Pain Scale) Improved compliance with treatment duration Reduced need for pain/anxiety medication Equivalent or better seal effectiveness Clinician acceptability (questionnaire score >4) Reduced nursing time by ≥20% Economic value through time and cost savings

At each dressing change and final removal, qualitative data from clinicians will assess the acceptability and usability of Comfort Release® NPWT drapes.

DETAILED DESCRIPTION:
Study Overview: Two-Aimed NPWT Drape Clinical Trial

Global Biomedical Technologies is advancing a novel surgical drape for negative pressure wound therapy (NPWT) that leverages Comfort Release®-a "switchable adhesive" technology designed for painless and trauma-free removal. This innovative adhesive incorporates oligo(glycerol sebacate) (OGS) and polyacrylate, allowing strong bonding during use and rapid release upon exposure to isopropyl alcohol (IPA). This product addresses the unmet need for effective NPWT adhesives that prevent medical adhesive-related skin injuries (MARSI) without compromising performance.

Key Features of Comfort Release® Adhesive:

* Composition: OGS, a biodegradable elastomer pre-polymer, forms hydrogen bonds with IPA, enabling adhesive release.
* Performance: A >70% drop in adhesive strength within 5 seconds of 70% IPA application.
* Benefits: Reduces pain and trauma at removal, maintains effective NPWT seals, and improves patient outcomes.

This Direct-to-Phase II study compares the Comfort Release® NPWT drape with the market leader, V.A.C. drape (KCI Technologies, Inc.), focusing on clinical performance, patient outcomes, and clinician feedback.

Study Objectives:

1. Evaluate Performance: Assess the skin irritation, pain, seal effectiveness, and clinician usability of the Comfort Release® drape.
2. Provide Clinical Validation: Gather data for FDA 510(k) clearance, supporting the introduction of a novel NPWT adhesive drape to the market.

   Purpose:

   NPWT is commonly used for the management of more than 100 indications, including chronic wounds, acute open wounds, burns, and post operative sites. An estimated 6.5 million patients suffer from chronic wounds and an estimated 48 million inpatient surgeries are performed each year in the US3,4. NPWT involves covering a wound with an airtight dressing, sealed by adhesive, and applying sub-atmospheric pressure via a vacuum device. Strong adhesives are typically required for NPWT drapes. Exudate can leak with weaker adhesives, tainting peri-wound skin, causing loss of drape adherence, subsequently leading to the potential for macerated tissue, increased wound size, and slower or reduced healing. However, strong adhesives substantially increase the risk for medical adhesive-associated skin injuries (MARSI) during drape removal/changes. Drape removal can cause epidermal layers to separate and/or detach from the dermis, resulting in skin tears and moisture-associated skin damage, and skin irritation. Studies show the type of drape used correlates with acute pain during dressing changes and injury to the peri-wound tissue, in turn delaying the wound healing process. Previous attempts to develop a product with strong adhesion and easy removability have fallen short. Silicone adhesives have poor skin adherence and are expensive, thus requiring stronger adhering acrylic sealing strips or other acrylic components to mitigate leaks. Addressing this unmet need, Global Biomedical Technologies has developed an adhesive acrylic NPWT drape incorporating innovative ester oligomers that release from the skin with the addition of isopropyl alcohol. This painless adhesive technology, "Comfort Release®," has proven high patient satisfaction with low incidence of MARSI. This project will confirm the superior functionality and acceptability of Comport Release® NPWT drapes against the market leader (V.A.C. drape by KCI Technologies, Inc.) in both single-use and serial-use NPWT applications. The data obtained from this Direct to Phase II project is expected to support a 510K FDA clearance.

   The proposed research aims to provide the clinical validation and data needed for a510K FDA clearance. If successful, the knowledge gained as a result of this trial can bring to market a novel surgical drape for wound therapy that has strong potential to be pain-free and atraumatic and will help facilitate wound healing. This can potentially contribute to improved patient outcomes. Given that there are minimal risks in this trial we find them reasonable to obtain the knowledge and clinical data needed bring this drape to pursue FDA clearance and bring this novel NPWT drape to market.

   Addressing this, Global Biomedical Technologies will compare Comfort Release® NPWT drape with an innovative "switchable adhesive" technology for painless and trauma free removal with the standard KCI V.A.C.® drape in post-surgical wound patients. The types of post-op wounds that receive NPWT that are eligible for this study include adult acute wounds and incisions, as well as chronic wounds and burns.

   ________________________________________

   Study Design:

   Single-Center, Two-Armed, Randomized Trial
   * Aim 1: Short-duration use (200 patients):

     o Assess single-use (in most cases) application, skin irritation, pain at removal, and seal effectiveness.
     * Study duration: Approximately 2 years.
     * Population: General post-surgical patients.
   * Aim 2: Serial-use application (100 patients):

     * Assess cumulative effects, including MARSI incidence, narcotic usage, compliance, and leak rates.
     * Study duration: Approximately 2 years.
     * Population: Chronic wound patients undergoing serial NPWT.

   Assessments:

   • Skin Irritation and Injury:
   * Tool: MARSI scoring system (erythema, tension blisters, maceration, etc.).
   * Immediate and 30-minute post-removal assessments.

     * Pain Evaluation:
   * Scale: Indiana Polyclinic Combined Pain Scale (0-10).

     • Seal Effectiveness:
   * Leak incidence recorded by clinicians.

     • Treatment Compliance:
   * Monitoring adherence to prescribed NPWT regimens.

     • Medication Use:
   * Tracking pain and stress-reducing medication usage.

     • Clinician Acceptability:
   * Documented via case report forms.

   Risk Mitigation and Ethical Considerations:

   • Minimal Risks:
   * Potential for skin irritation or discomfort, inherent to NPWT.
   * Breach of confidentiality mitigated through deidentification and secure data storage.

     • Informed Consent:
   * Lay-language consent forms provided, ensuring participants fully understand study procedures, risks, and benefits.
   * Oversight by Denise Anderson, RN, WCC, with site coordinators. • Adverse Event Reporting:
   * Immediate reporting of new risks or adverse events to the Columbia IRB.

   Statistical and Sample Size Justification:
   * Aim 1: 100 patients/group (200 total) across three sites (WCM, CUIMC, AMC). o Effect size: Moderate (d=0.4); significance at α=0.05 with 80% power.
   * Aim 2: 50 patients/group (100 total) at two sites (WCM, VMR). o Effect size: Moderate (d=0.6), targeting higher MARSI incidence in chronic cases.

   Sponsor & Principle-Investigator Howard S. Rosing, MD, PhD CEO, Global Biomedical Technologies, LLC 6350 Lake Oconee Pkwy, Ste 110, PMB 11 Greensboro, GA 30642 Contact: hrosing@comfortrelease.com Phone: (m) 239-330-5646 (o) 833-726-9269 Ext 710

   Principle-Investigator:

   Robert John Winchell, MD Chief, Division of Trauma & Burns Weill Cornell Medical Center (WCM) 525 East 68th Street, Room P7-714, Box 116 New York, NY 10065 Contact: row9057@med.cornell.edu Phone: 646-962-8490

   Co-Principle Investigator:

   Jarrod Terrence Bogue, MD Clinical Instructor in Surgery, Columbia University Urving Medical Center (CUIMC) 161 Fort Washington Avenues, Suite 5 New York, NY 10032 Contact: jb3892@cumc.columbia.edu Phone: 203-668-8595

   Co-Principle Investigator:

   Daniel Careage, MD- Careaga Plastic Surgery 220 Alhambra Circle, First Floor Coral Gables, FL 33134 Absolute Medical Center (AMC) 5040 Northwest 7th Street Suite 500 Miami, Florida 33126 Contact: Juan Diaz drdiaz@absolutemedicalcenter.com> 305-508-0004

   Co-Principle Investigator:

   Deeza Frankel, DPM Vital Medical Research (VMR) 10780 W Flagler ST, Suite #6 Sweetwater, FL 33174 Contact: Alejandro Morlan, APRN Alejandro.m@vitalmedicalresearch.com 305-703-4414

   IRB Compliance: Advarra IRB serves as the single IRB for all participating sites. Advarra IRB is fully accredited by the Association for the Accreditation of Human Research Protection Programs (AAHRPP).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older post-surgical inpatients with a plan of treatment using NPWT
2. Able to communicate and consent to participation in the study
3. Access to V.A.C. by KCI drape and NPWT kits
4. Able to report pain level using a pain scale.
5. If outpatient- able to return to the clinic for all drape/dressing changes

Exclusion Criteria:

1. History of known hypersensitivity to acrylic adhesives
2. History of known hypersensitivity to isopropyl alcohol
3. The patient is expected to be unconscious during the drape removal/change
4. Under the age of 18 years 5. Unable to give consent, including language barrier, unless an interpreter is readily available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Medical Adhesive-Related Skin Injury (MARSI). | From the first drape removal to the end of treatment- 1 to 8 weeks.
  Measure: The percentage of patients experiencing Medical Adhesive-Related Skin Injury from surgical drape removal as assessed using the MARSI scale upon drape removal, and, if any abnormality is noted, a second MARSI assessment is completed. If there is a MARSI score of 1 or 2 = follow up assessment in completed in approximately 15 minutes, and a score of 3 or 4 = follow up assessment is completed in approximately 30 minutes.
Patient-reported pain scores during drape removal. | From enrollment to the end of treatment - from 1 - 8 weeks.
  Pain intensity scored on the Indiana Polyclinic Combined Pain Scale during the drape removal. Scale of 0 to10, 0 = no pain and 10= worst imaginable pain.
Change in medication use for anxiety, pain, and stress. | From enrollment to the end of treatment - from 1 - 8 weeks.
  Measure: Quantity (e.g., dosage or frequency) of medications used for anxiety, pain, and stress related to drape removal.
Drape seal integrity (leak incidence rate). | From enrollment to the end of treatment - from 1 - 8 weeks.
  Proportion of drapes maintaining an effective seal compared to or the control drape.
Patient drop-out rate from NPWT treatment due to drape issues. | From enrollment to the end of treatment - from 1 - 8 weeks.
  Measurement: Percentage of patient who discontinue NPWT treatment before completing the prescribed treatment duration drop-out from the prescribed treatment duration to determine how much pain and skin injury plays a role in patient compliance.

SECONDARY OUTCOMES:
Clinician Acceptability of Comfort Release® drape. | From application of the first drape to the end of treatment - from 1 - 8 weeks.
  Measure: Time taken by the clinician (in minutes) to remove the NPWT drape while minimizing the pain the patient suffers from the drape removal. This time-saving measurement could increase the economic value of the drape.

CONTACTS AND LOCATIONS:
Overall Officials: Howard S Rosing, MD, PhD, Principal Investigator — Global Biomedical Technologies, LLC
Locations (4):
- United States (4):
  - Absolute Medical Center, LLC, Miami, Florida
  - Vital Medical Research, Sweetwater, Florida
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Study patient results within the 2 Aims against the control - market leader product results.
Supporting Information: Study Protocol, ICF
Time Frame: Jan 6, 2025
Access Criteria: Health care professional status is required. All requests for access will be emailed to danderson@comfortrelease.com.

REFERENCES:
- [Background] The Indiana Polyclinic Combined Pain Scale. 2022. at https://www.painscale.com/article/the - indiana -polyclinic- combined - pain - scale .)
- [Background] McNichol L, Lund C, Rosen T, Gray M. Medical adhesives and patient safety: state of the science: consensus statements for the assessment, prevention, and treatment of adhesive-related skin injuries. J Wound Ostomy Continence Nurs. 2013 Jul-Aug;40(4):365-80; quiz E1-2. doi: 10.1097/WON.0b013e3182995516. PMID 23759927
- [Background] Negative Pressure Wound Therapy Market Size, Share & Trends Analysis Report By Product (Conventional NPWT, Single- use NPWT), By Wound Type (Diabetic Foot Ulcers, Venous Leg Ulcers), By End Use, By Region, And Segment Forecasts, 2022 - 2030. 2022. (Accessed July 18, 2022, at https://www.grandviewresearch.com/industry - analysis/negative - pressure - wound - therapy - npwt - market .
- [Background] Fumarola S, Allaway R, Callaghan R, Collier M, Downie F, Geraghty J, Kiernan S, Spratt F, Bianchi J, Bethell E, Downe A, Griffin J, Hughes M, King B, LeBlanc K, Savine L, Stubbs N, Voegeli D. Overlooked and underestimated: medical adhesive-related skin injuries. J Wound Care. 2020 Mar 1;29(Sup3c):S1-S24. doi: 10.12968/jowc.2020.29.Sup3c.S1. No abstract available. PMID 32134695
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] National Health Statistic Report, Number 102, February 28, 2017
- [Background] Apelqvist J, Willy C, Fagerdahl AM, Fraccalvieri M, Malmsjo M, Piaggesi A, Probst A, Vowden P. EWMA Document: Negative Pressure Wound Therapy. J Wound Care. 2017 Mar 1;26(Sup3):S1-S154. doi: 10.12968/jowc.2017.26.Sup3.S1. PMID 28345371
- [Background] Zaver V, Kankanalu P. Negative Pressure Wound Therapy. 2023 Sep 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK576388/ PMID 35015413
- [Background] Robertson F, Wang Y, Rosing H. An oligomeric switch that rapidly decreases t he peel strength of a pressure-sensitive adhesive. International Journal of Adhesion and Adhesives 2014; 55:64-8
- [Background] Upton D, Solowiej K, Hender C, Woodyatt KY. Stress and pain associated with dressing change in patients with chronic wounds. J Wound Care. 2012 Feb;21(2):53-4, 56,58 passim. doi: 10.12968/jowc.2012.21.2.53. PMID 22584524
- [Background] Upton D, Andrews A. Pain and trauma in negative pressure wound therapy: a review. Int Wound J. 2015 Feb;12(1):100-5. doi: 10.1111/iwj.12059. Epub 2013 Mar 12. PMID 23489350
- [Background] Vuerstaek JD, Vainas T, Wuite J, Nelemans P, Neumann MH, Veraart JC. State-of-the-art treatment of chronic leg ulcers: A randomized controlled trial comparing vacuum-assisted closure (V.A.C.) with modern wound dressings. J Vasc Surg. 2006 Nov;44(5):1029-37; discussion 1038. doi: 10.1016/j.jvs.2006.07.030. Epub 2006 Sep 26. PMID 17000077
- [Background] Wang Y, Ameer GA, Sheppard BJ, Langer R. A tough biodegradable elastomer. Nat Biotechnol. 2002 Jun;20(6):602-6. doi: 10.1038/nbt0602-602. PMID 12042865
- See also: Comfort Release® website. — https://comfortrelease.com/

DOCUMENTS (3):
  • Study Protocol (2025-10-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT06717308/Prot_007.pdf
  • Statistical Analysis Plan (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT06717308/SAP_005.pdf
  • Informed Consent Form (2025-11-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT06717308/ICF_008.pdf